CLINICAL TRIAL: NCT00729898
Title: Safety of NovoMix® 30 (Biphasic Insulin Aspart) Treatment in Patients With Type 2 Diabetes
Brief Title: Observational Study to Observe the Safety of NovoMix® 30 Treatment in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3512
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoMix® 30

SUMMARY:
This study is conducted in Europe. The study aims to observe the incidence of serious adverse drug reactions in patients with type 2 diabetes during NovoMix® 30 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with diabetes type 2 diabetes
* Currently treated with basal human insulin therapy (basal only or in combination with oral glucose lowering drugs or other insulin
* Selection of patients will be at the discretion of the treating physician after the decision to prescribe one of the study products to the patient

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Pregnancy, breast-feeding or intention of becoming pregnant within the next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population type 2 diabetes strated on NovoMix® 30
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions, including major hypoglycaemic events | after 12 and 26 weeks

SECONDARY OUTCOMES:
Number of all hypoglycaemic events | in the 4 weeks preceding visit, at 12 weeks and the final visit at 26 weeks
Number of all adverse drug reactions | after 12 and 26 weeks
HbA1c | at 12 and 26 weeks
Variability in fasting plasma glucose (FPG) values and average FPG levels | at visits at 12 and 26 weeks
Weight changes | at visits at 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Rud, Norway
- Novo Nordisk Investigational Site, Farsta, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com